CLINICAL TRIAL: NCT07079488
Title: Motor Development in Infants and Toddlers Affected by Vestibular Impairment
Brief Title: Vestibular Function and Motor Development in Small Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Luca Verrecchia, Principal Investigator, Region Stockholm
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: K2023-7366
Record Dates: First submitted 2023-10-12; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vestibular impairment (Other)
  Interventions: Diagnostic Test: Motor proficiency scales
- control subject (Other)
  Interventions: Diagnostic Test: Motor proficiency scales

INTERVENTIONS:
Diagnostic Test: Motor proficiency scales — AIMS, PDMS-2, HINE

SUMMARY:
Infants and toddlers with and without vestibular impairment will be tested blinded by pediatric physiotherapist with different age adequate motor scales in order to find out pathological motor patterns specifically associated to vestibular impairment.

ELIGIBILITY:
Inclusion Criteria:

vestibular impairment normal vestibular function -

Exclusion Criteria:

children unable to be tested with chield-friendly vestibular testing

-

Ages: 5 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales II | at enrollment and at 6 months
  Pathological motor patterns
Alberta Infant Motor Scales | at enrollment and at 6 months
  Pathological motor patterns
Hammersmith Infant Neurological Examination checklist | at enrollment and at 6 months
  Pathological motor patterns

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Univerisity Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided